CLINICAL TRIAL: NCT02585427
Title: Effects of Co-ingesting a Low/High GI Meal With Different Fat Saturation on Postprandial Glucose, Insulin, and Triacylglycerol Responses in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/00719
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Diabetes; Obesity; metabolic disorders
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Metabolic Diseases | interventions — Butter; Olive Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- low glycemic index rice with butter (Experimental): 50 g available low glycemic index rice cooked with 48 g butter ( equal 40 g saturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil
- low glycemic index rice with olive oil (Experimental): 50 g available low glycemic index rice cooked with 44 g olive oil ( equal 40 g monounsaturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil
- low glycemic index rice with grapeseed oil (Experimental): 50 g available low glycemic index rice cooked with 40 g grapeseed oil ( equal 40 g polyunsaturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil
- high glycemic index rice with butter (Experimental): 50 g available high glycemic index rice cooked with 48 g butter ( equal 40 g saturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil
- high glycemic index rice with olive oil (Experimental): 50 g available high glycemic index rice cooked with 44 g olive oil ( equal 40 g monounsaturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil
- high glycemic index rice with grapeseed oil (Experimental): 50 g available high glycemic index rice cooked with 40 g grapeseed oil ( equal 40 g polyunsaturated fatty acid)
  Interventions: Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil

INTERVENTIONS:
Dietary Supplement: low glycemic index rice, high glycemic index rice, butter, olive oil and grapeseed oil

SUMMARY:
It is now recognized that diet plays a critical role in the etiology and management of the chronic diseases such as diabetes, obesity and cardiovascular disease. A high consumption of fat, especially saturated fat, is an established risk factor for Cardiovascular Disease.The glycaemic index (GI) is a measurement of the ability of different types of carbohydrate-based foods to raise blood glucose. The interest in low GI food as a weight management tool has been increasing. Different types of carbohydrates differ in their ability to increase postprandial blood glucose and insulin secretion, and may also modulate the effect of different fatty acids. The current study will compare the consumption of low and high GI carbohydrate with different fat saturation on postprandial glucose, insulin, and triacylglycerol responses in healthy participants.

The data generated will have direct applications in public health policy and clinical nutrition management of chronic disease. The outcomes of the study will significantly contribute to the long term national goals of Singapore to manage and to reduce the incidence of chronic disease associated with the metabolic syndrome.

DETAILED DESCRIPTION:
This study will be conducted using a randomized, crossover design with six dietary phases: a low GI meal or a high GI meal with saturated fat, monounsaturated fat or polyunsaturated fat. All participants will be randomly allocated to the six test meals, with the order balanced. Fifteen participants aged between 21 and 40 years will be recruited from the general public in Singapore. During the testing session, a maximum of eleven blood samples will be collected by fingerpricks and cannulation. Fingerpricks and cannulation may cause minor discomfort and there may be some slight bruising around the site. Fingerpricks and cannulation will be done by an experienced research nurse or a trained research officer to minimize participant discomfort. If bruising does occur, it should disappear within one day and it should not affect participants' regular daily activity. Participants will be limited to a maximum of two tests per week. In addition, blood collection will be carried out in a sterile designated area and thus the risk of infection will be very low. On rare occasions, participants may feel unwell during or after the testing session. The investigators have several metabolic suites with beds for these individuals to rest on. The research nurse and research officers will monitor the individuals' condition and they will be provided with a ride home if required.

All the study foods will be prepared in a hygienic manner in a purpose-built research kitchen maintained to the highest hygiene standards. The research staff has undergone basic training in food hygiene procedures. Hence, the risk of infective acute gastroenteritis will be minimal.

A number of dietary interventions have aimed to investigate the effect of dietary fat quality on glucose, insulin and lipidemia response. Up to now there have been few studies connect the glycaemic load and fat quality together. The investigators study's results will help public choose fat quality and carbohydrate quality in the diet. Participants will be provided with some snacks at the end of each testing session.

In addition, participants will be provided with their blood glucose, blood insulin, blood lipid profile, blood pressure, and body composition results, with a brief interpretation of these at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male subjects aged between 21 and 40 years
* Do not have major chronic disease such as heart disease, cancer or diabetes mellitus
* Do not have family history of diabetes
* Do not have intolerances or allergies to test products(wheat and milk based products)
* Not taking insulin or drugs known to affect glucose or triglyceride levels and body fat distribution
* Do not have major medical or surgical event requiring hospitalization within the preceding three months

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Glucose response of different treatments | 4 hours postprandial
  The blood glucose will be measured by finger prick and venous blood collection at the same time points
Insulin response of different treatments | 4 hours postprandial
  Insulin concentration will be measured by COBAS Roche analyzer e311
Triglycerides response of different treatments | 4 hours postprandial
  Triglycerides will be measured by COBAS Roche analyzer e411

SECONDARY OUTCOMES:
Active Glucagon-like peptide 1 response of different treatments | 4 hours postprandial
  Active Glucagon-like peptide 1 will be measured by Multiplex kits
Gastric inhibitory polypeptide response of different treatments | 4 hours postprandial
  Gastric inhibitory polypeptide will be measured by Multiplex kits

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore

REFERENCES:
- [Derived] Sun L, Tan KWJ, Lim JZ, Magkos F, Henry CJ. Dietary fat and carbohydrate quality have independent effects on postprandial glucose and lipid responses. Eur J Nutr. 2018 Feb;57(1):243-250. doi: 10.1007/s00394-016-1313-y. Epub 2016 Oct 21. PMID 27770188